CLINICAL TRIAL: NCT07047352
Title: A Multi-center Single Arm Prospective Study in Patients of Hematological Malignancies Colonized With Carbapenem-resistant Bacterials to Evaluate the Timing of Empirical Antibiotic Treatment (CROEAT Study)
Brief Title: Prospective Study Evaluate the Timing of Empirical Treatment for Carbapenem-resistant Bacterials (CROEAT Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-BMT-2403
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Carbapenem-resistant Enterobacterales; Neutropenia; Hematological Malignancies
Keywords: carbapenem-resistant enterobacterales; hematological malignancies; neutropenia; empirical therapy
MeSH Terms: conditions — Neutropenia; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Empirical antibiotics treatment covering carbapenem-resistant enterobacterales (CRE) in neutropenic patients with positive CRE colonization after screening to meet the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study: empirical treatment (Experimental): Empirical treatment to cover carbapenem-resistant enterobacterales
  Interventions: Other: Empirical treatment

INTERVENTIONS:
Other: Empirical treatment — Empirical treatment to cover carbapenem-resistant enterobacterales

SUMMARY:
In this study, we will evaluate the feasibility and clinical outcomes of risk adaptive empirical therapy to cover carbapenem resistance gram negative bacteria (CRO) in patients with hematological malignancies colonized with CRO. Patients assessed by the clinician as being at high risk for CRO infection and requiring intravenous antibiotics covering CRO must meet the following conditions:

1. Positive active screening for CRO or past CRO infection or local prevalence of CRO (e.g.,CRO detection rate>20% among recently hospitalized patients);
2. Presence of fever or other possible signs and symptoms of infection;
3. Neutropenia(ANC<0.1×10^9/L)expected to last for ≥7 days,and having any of the following:

   * Gastrointestinal mucositis/peri-anal infection/intestinal obstruction;

     * Shock or severe sepsis;

       * Respiratory failure:deoxygenated PaO2<60 mmHg or requiring mechanical ventilation;

         * Disseminated intravascular coagulation;

           * Altered mental status or psychiatric abnormalities;

             * Congestive heart failure requiring treatment;

               * Arrhythmia requiring treatment;

                 * Recurrence of fever shortly after cessation of or during empirical treatment with carbapenems (≤7 days).

The endpoints of study include incidence of blood-stream infection by CRO, incidence of all causes mortality, incidences of clinical and microbiology response.

DETAILED DESCRIPTION:
Neutropenic fever is common in patients with hematological malignancies undergoing chemotherapy or transplantation. Empirical antibiotics therapy is essential treatment principle. In China, recent evidence demonstrated that the carbapenem resistant gram negative bacteria was emerging as an important issue and CRO colonization was positive in about 10% of patients by rectal swab. In such group of patients, the empirical treatment of patients with neutropenic fever therapy remained as a challenge. In this study, we plan to evaluate the feasibility and clinical outcomes of risk adaptive empirical therapy to cover CRO in patients with hematological malignancies colonized with CRO.

Patients assessed by the clinician as being at high risk for CRO infection and requiring intravenous antibiotics covering CRO must meet the following conditions:

1. Positive active screening for CRO or past CRO infection or local prevalence of CRO (e.g.,CRO detection rate>20% among recently hospitalized patients);
2. Presence of fever or other possible signs and symptoms of infection;
3. Neutropenia(ANC<0.1×10^9/L)expected to last for ≥7 days,and having any of the following:

   * Gastrointestinal mucositis/peri-anal infection/intestinal obstruction;

     * Shock or severe sepsis;

       * Respiratory failure:deoxygenated PaO2<60 mmHg or requiring mechanical ventilation;

         * Disseminated intravascular coagulation;

           * Altered mental status or psychiatric abnormalities;

             * Congestive heart failure requiring treatment;

               * Arrhythmia requiring treatment;

                 * Recurrence of fever shortly after cessation of or during empirical treatment with carbapenems (≤7 days).

The endpoints of study include incidence of blood-stream infection by CRO, incidence of all causes mortality, incidences of clinical and microbiology response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies receiving hospital treatment such as chemotherapy/immunotherapy/hematopoietic stem cell transplantation;
* Those with a recent history of CRO colonization or who have been screened for CRO once a week continuously since admission;
* Patients assessed by the clinician as being at high risk for CRO infection and requiring intravenous antibiotics covering CRO must meet the following conditions:

  1. Positive active screening for CRO or past CRO infection or local prevalence of CRO (e.g.,CRO detection rate>20% among recently hospitalized patients);
  2. Presence of fever or other possible signs and symptoms of infection;
  3. Neutropenia(ANC<0.1×10^9/L)expected to last for ≥7 days,and having any of the following:

     * Gastrointestinal mucositis/peri-anal infection/intestinal obstruction;

       * Shock or severe sepsis;

         * Respiratory failure:deoxygenated PaO2<60 mmHg or requiring mechanical ventilation;

           * Disseminated intravascular coagulation;

             * Altered mental status or psychiatric abnormalities;

               * Congestive heart failure requiring treatment;

                 * Arrhythmia requiring treatment;

                   * Recurrence of fever shortly after cessation of or during empirical treatment with carbapenems (≤7 days).
* The patient or their legal guardian has signed the informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Individuals who are expected to die within 14 days of hospitalization or have an expected hospital stay of less than 7 days;
* Any conditions that the investigator believes may increase the risk to the patient;
* Severe psychological or psychiatric disorders with poor estimated compliance;
* The presence of any other conditions that the investigator deems unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of overall mortality | 14 days
  Patients died of any causes

SECONDARY OUTCOMES:
Incidence of documented CRE blood stream infection | 30 days
  Patients with positive culture of carbapenem-resistant enterobacterales
Clinical response | 14 days
  Patients with full recovery of clinical signs and symptoms of infection
microbiology response | 14 days
  Patients with clearance of blood carbapenem-resistant enterobacterales

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, Principal Investigator — Ruijin Hospital
Locations (1):
- Rui Jin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No